CLINICAL TRIAL: NCT04483908
Title: COVID-19 in Baselland: Investigation and Validation of Serological Diagnostic Assays and Epidemiological Study of Sars-CoV-2 Specific Antibody Responses (SERO-BL-COVID-19)
Brief Title: COVID-19 in Baselland: Investigation and Validation of Serological Diagnostic Assays and Epidemiological Study of Sars-CoV-2 Specific Antibody Responses
Acronym: SEROBL-COVID19
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETH Zurich (Switzerland) (Other); Health Department of the Canton of Basel-Stadt (Other Government)
Responsible Party: Sponsor
Other Study IDs: BASEC Project-ID 2020-00816
Record Dates: First submitted 2020-07-22; First posted 2020-07-23 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Infection
Keywords: Sars-CoV-2 infection; ELISA test; lateral flow assay; point of care (POC) assay; saliva based serology
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Immune cells (B cells and T cells) from peripheral blood mononuclear cells (PBMC) from the cohort of COVID-19 recovered patients will be subjected to bulk and single-cell RNA sequencing (RNA-seq). Biological material in this project is not identified by participant name but by a unique participant number. Biological material is appropriately stored in a restricted area only accessible to authorized personnel. Biobank is handled by the accredited diagnostic lab of the Swiss TPH according to the rules of clinical sample storage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Disease survivors with a positive polymerase chain reaction (PCR) test > 12days (d) ago and no symptoms (~250 participants).
  Cohort 1 & 2 are supposed to have an antibody response to different levels and should provide ability to deduce the detection limit, and estimate the true positive and false negative rates of both ELISA and POC assays.
  Interventions: Diagnostic Test: blood draw; Diagnostic Test: fingertip tests for POC assays; Diagnostic Test: saliva collection
- Cohort 2: Disease survivors with a positive PCR test 7 - 12d ago and no symptoms (~100 participants).
  Cohort 1 & 2 are supposed to have an antibody response to different levels and should provide ability to deduce the detection limit, and estimate the true positive and false negative rates of both ELISA and POC assays.
  Interventions: Diagnostic Test: blood draw; Diagnostic Test: fingertip tests for POC assays; Diagnostic Test: saliva collection
- Cohort 3: Subjects with PCR negative test > 5d (~100 participants). Cohort 3 & 4 are the control groups. They are supposed to not have an antibody response for COVID-19 and should therefore help estimate the true negative and false positive rates.
  Interventions: Diagnostic Test: blood draw; Diagnostic Test: fingertip tests for POC assays; Diagnostic Test: saliva collection; Diagnostic Test: collection of swabs
- Cohort 4: Anonymised blood sera from the "Serumbank" at the Kantonsspital Basel-Land (KSBL) taken during last years influenza period (~100 participants).
  Cohort 3 & 4 are the control groups. They are supposed to not have an antibody response for COVID-19 and should therefore help estimate the true negative and false positive rates.
  Interventions: Diagnostic Test: blood draw

INTERVENTIONS:
Diagnostic Test: blood draw — 2x 10ml of blood, one vial to obtain the antibodies and one vial in ethylenediaminetetraacetic acid (EDTA) (or citrate-treated) to obtain peripheral blood mononuclear cells (PBMCs)
Diagnostic Test: fingertip tests for POC assays — performing POC test by taking two blood drops from the fingertip
  Groups: Cohort 1; Cohort 2; Cohort 3
Diagnostic Test: saliva collection — saliva collection: the patient delivers saliva into an adsorbent filter, which is placed in the Salivette tube, centrifuged at 1,600x g for 15 min at 4°C to remove cells and debris. Native supernatant is used for testing.
  Groups: Cohort 1; Cohort 2; Cohort 3
Diagnostic Test: collection of swabs — collection of nasopharyngeal and oropharyngeal swabs for PCR testing on the control group (eg negative subpopulation)
  Groups: Cohort 3

SUMMARY:
The study is to investigate the antibody response in the blood and saliva of people with a known COVID-19 infection in the canton of Baselland.

DETAILED DESCRIPTION:
This study is to analyse the antibody response in the blood and saliva of people with a known COVID-19 infection in the canton of Baselland.

The study aims to validate strategies to measure antibody levels with minimal intervention and to explore the antibody response and technical capacity for said measurement. The study will collect the minimally necessary samples to deduce a strategy for serum or saliva surveillance of the population of the canton Baselland. To achieve this, the study is designed to address the following points:

* determine specificity, sensitivity and general utility of point of care (POC) and ELISA tests to deduce a strategy for serum surveillance of the population of the canton Baselland
* especially validate different POC kits in regard of their use for continuous surveillance
* gain an understanding of seroconversion and antibody levels of patients and survivors
* gain an understanding of the individual antibody and T-cell repertoire of patients and survivors
* study whether patterns of convergent antibody evolution is generated in the surviving population or whether the diseases survivors generated an antibody pool recognizing a specific epitope
* develop the technology to correlate blood antibody levels with levels detected in the saliva
* develop high throughput technologies for the precise detection of immune cell Repertoire and binding epitopes

ELIGIBILITY:
Inclusion Criteria:

* tested positive for COVID-19 in Baselland
* tested negative for COVID-19 in Baselland. Specifically, needed to show symptoms to be able to deduce cross reactivities.

Exclusion Criteria:

* continuous steroid therapy / chemotherapy / immunsuppressiva
* subject is treated for cancer
* severe autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from the database of all positive PCR cases for COVID-19 tested in the canton Basel-Land.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Qualitative method validation (yes/ no) | at baseline
  Qualitative method validation: qualitative result of the ELISA (Patient does / does not have immunity) as the gold standard compared to the POC using univariate measures to derive sensitivity and specificity of the POC.
Quantitative method validation (antibody concentrations) | at baseline
  Quantitative method validation: antibody concentration from the ELISA are related to the dichotomous result from POC.

SECONDARY OUTCOMES:
Immune cell repertoire sequencing | at baseline
  Antibody and T cell repertoires and transcriptional profiles of cells will be used to identify potential antibody and T cell clones correlated with COVID-19 protection.

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Savic, Dr. med., Principal Investigator — Department of Health, Economics and Health Directorate Canton Basel-Land
Locations (1):
- Department of Health, Economics and Health Directorate Canton Basel-Land, Liestal, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The Biobank data is planned to be shared according to the Biobank regulatory approved by the EKNZ